CLINICAL TRIAL: NCT06581757
Title: Evaluation of the Predictive Value of Serum Glial Fibrillary Acidic Protein and Ubiquitin Carboxy-terminal Hydrolase L1 for Subarachnoid Haemorrhage
Brief Title: Serum GFAP and UCHL1: Evaluation of Their Predictive Value for SAH
Acronym: SAH
Status: Terminated | Type: Observational
Why Stopped: The study has been terminated as the team did not have the amount of positives they were expecting and the CI has got early employment at another Trust and will not be carrying on the project.
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024LAB134
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Subarachnoid Haemorrhage (SAH)
Keywords: Subarachnoid haemorrhage; Evaluation; SAH; Glial Fibrillary Acidic Protein; Ubiquitin Carboxy-terminal Hydrolase L1; Cerebrospinal Fluid; Lumbar Puncture
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The study will utilise residual, surplus serum samples that have already been taken as part of the patient's routine care. The patients have already been consented for investigation of SAH and the leftover sample would otherwise be discarded by the laboratory.
  Samples will be identified by the co-investigator, whom is part of the normal clinical care team, using a data gather from the pathology laboratory information management system of patients that have had a serum sample taken within 24 hours of a test for CSF xanthochromia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residual, surplus serum samples: The study will utilise residual, surplus serum samples with a minimum volume of 300µl that have already been taken as part of the patient's routine care. The patients have already been consented for investigation of SAH and the leftover sample would otherwise be discarded by the laboratory.

SUMMARY:
To verify the analytical performance of GFAP and UCH-L1 biomarkers marketed by Abbott Diagnostics and to assess diagnostic accuracy of these biomarkers in predicting subarachnoid haemorrhage

DETAILED DESCRIPTION:
Subarachnoid haemorrhage (SAH) refers to blood entering the subarachnoid space and may be due to aneurysmal or non-aneurysmal causes. Patients with SAH characteristically present with a sudden onset 'thunderclap' headache (Patel et al., 2021). This is an acute medical emergency and is the third most common type of stroke, with approximately 500,000 cases annually across the world (Claassen and Park, 2022). Morbidity has decreased over the past few decades, however, there is still an approximate 35% occurrence of death within three months of a SAH (Andersen et al., 2019). Early diagnosis is important to enable timely treatment and thereby improve prognosis. Current NICE guideline NG228 state the diagnosis of SAH is to be made from a non-contrast CT scan showing the presence of blood in the subarachnoid space. A negative CT done within 6 hours of symptom onset is considered not indicative of a SAH. If however, the CT is 'negative' and is performed more than 6 hours after onset of symptoms then a LP is advised to look for the presence of xanthochromia in the CSF (NICE, 2022).

Xanthochromia refers to the yellowing of the cerebrospinal fluid (CSF) due to accumulation of bilirubin from the breakdown of red blood cells in the subarachnoid space. Its presence, in the appropriate clinical context, confirms a diagnosis of SAH. In our population, approximately 10% of CSF xanthochromia tests confirm SAH, meaning 90% of LPs may not have been necessary. This test is reliable only if performed at least 12 hours after the onset of symptoms. The xanthochromia test is considered a manual test and requires trained and competent staff. There are multiple pre-analytical requirements in order to produce a reliable result. For example, the sample must be protected from light during transport and not transported by the air tube. Exposure to light can cause the bilirubin to breakdown which can then lead to a false negative result (Cruickshank et al., 2008). Samples transported in the pneumatic tube system may give false results due to the lysis of red cells.

Traumatic tap, in which the needle causes blood to enter the subarachnoid space, and which will then be present in the CSF sample can also cause interference as discolouration of the sample may mask xanthochromia. The least bloodstained CSF sample must therefore be used for analysis. Finally, an LP is an invasive procedure and is therefore an unpleasant experience for the patient (Long et al., 2017).

In summary, a test for SAH that is subject to fewer pre-analytical and analytical interferences would be superior to the current CSF xanthochromia test. Whilst it is not expected that a serum test could replace the need for CSF xanthochromia completely, a test that could identify which patients are likely to have negative LP could reduce the number of unnecessary LPs.

There are two candidate biomarkers - Ubiquitin C-terminal hydroxylase-L1 (UCH-L1) and Glial Fibrillary Acidic Protein (GFAP) - which have been found to increase in blood following brain damage and in traumatic brain injuries, including SAH. However, current guidelines (NICE, 2022) for SAH state that brain biomarkers are not currently recommended by guidelines as part of the SAH diagnosis pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old, who have had an LP with a serum sample taken within 24 hours of the LP.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to hospitals covered by the black country pathology service (BCPS) who have had a lumbar puncture (LP) for the investigation of subarachnoid haemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Measures of diagnostic accuracy including sensitivity, specificity, negative predictive value and positive predictive value. | 1 year
  Metrics of diagnostic accuracy to include sensitivity, specificity, negative predictive value and positive predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Young, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- New Cross Hospital, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No